CLINICAL TRIAL: NCT03140111
Title: Post-approval Study to Assess the Effectiveness of LAMELLEYE vs Comparator for the Treatment of Dry Eye Symptoms in Patients With Primary Sjögren's Syndrome
Brief Title: LAMELLEYE for the Treatment of Dry Eye Symptoms in pSS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Lamellar Biomedical Ltd (Industry); Robertson Centre for Biostatistics - University of Glasgow (Unknown); Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GN16HS410; 001172 (Other Grant/Funding Number: Lamellar Biomedical Ltd.)
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Dry Eye Syndromes; Primary Sjögren Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A, followed by Treatment B (Other): Treatment group that will receive Treatment A for 28 days, followed by Treatment B for 28 days. There will be a minimum 7 day washout between Treatments. LAMELLEYE Dry Eye Drops and OPTIVE FUSION will be administered to all subjects in this arm. Treatments will be self-administered at least 3 times a day.
  Interventions: Device: LAMELLEYE; Device: OPTIVE FUSION
- Treatment B, followed by Treatment A (Other): Treatment group that will receive Treatment B for 28 days, followed by Treatment A for 28 days. There will be a minimum 7 day washout between Treatments. LAMELLEYE Dry Eye Drops and OPTIVE FUSION will be administered to all subjects in this arm. Treatments will be self-administered at least 3 times a day.
  Interventions: Device: LAMELLEYE; Device: OPTIVE FUSION

INTERVENTIONS:
Device: LAMELLEYE — Liposomal multi-dose preservative-free sterile suspension which contains soy lecithin phospholipids, sphingomyelin and cholesterol, suspended in saline.
  Other Names: CXB/1-14
Device: OPTIVE FUSION — Multi-dose sterile solution which contains sodium hyaluronate 0.1%, sodium carboxymethylcellulose 0.5%, glycerine 0.9%, erythritol, boric acid, sodium citrate dihydrate, potassium chloride, calcium chloride dihydrate, magnesium chloride hexahydrate, and is preserved with PURITE® 0.01% which breaks down into natural tear components on the eye.

SUMMARY:
Single-blind, randomised, single centre, 2-way crossover pilot study to investigate the effectiveness of LAMELLEYE for the treatment of dry eye symptoms in patients with primary Sjögren's Syndrome.

DETAILED DESCRIPTION:
The study is a 2-way crossover design comprising 2 treatments: the CE-marked LAMELLEYE dry eye drops, and a CE-marked comparator product. All Participants will be allocated to a treatment group in a random order.

The study design allows observations to be made between the treatments at both an intra- and inter-patient level regarding relationships between the patient's disease specific quality of life, symptoms and adverse events, and satisfaction with treatments.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each Participant must meet each of the following:

1. Male or female aged ≥ 18 years and ≤ 79 years at date of consent
2. Primary Sjögren's Syndrome diagnosed by a rheumatologist
3. Patient has symptoms of dry eye, and has failed to achieve symptom relief on adequate trial of standard topical therapy
4. Willing and able to attend Glasgow Caledonian University Vision Sciences Eye Clinic for therapy assessment; and to comply with all procedures and follow-up visits
5. Participant must have personally given written informed consent to allow anonymised data to be used in publications and presentations.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria are met:

1. Females who are pregnant, planning pregnancy or breastfeeding
2. Active ocular infection or current corneal ulceration
3. Ocular surgery within 6 months of study start date
4. Current contact lens wear
5. Any prior and/or current topical ophthalmic treatments that in the opinion of the CI or PI may interfere with the study outcomes
6. Started or changed the dose of chronic systemic medication known to affect tear production including, but not limited to antihistamines, anticholinergics, antidepressants, diuretics, corticosteroids or immunomodulators within 30 days prior to enrolment
7. Participants with known allergies to ingredients in any of the study treatments, or fluorescein
8. Participants who are judged inappropriate for inclusion in the study by the CI or PI.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-10-16 (Estimated); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Patient reported symptoms | 28 days (analysed for each treatment period)
  Ocular Surface Disease Index (OSDI):
  12-item questionnaire designed to assess the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning
  and Symptom Assessment in Dry Eye (SANDE): Two questions which each use a horizontal visual analogue technique to quantify patient symptomatology of dryness and/or irritation
Patient reported quality of life | 28 days (analysed for each treatment period)
  Impact of Dry Eye Disease on Everyday Life (IDEEL - copyright Novartis Pharma AG):
  The use of this questionnaire (Treatment Satisfaction module only) will provide assessment of the impact of study treatment on patient outcomes in this study.

SECONDARY OUTCOMES:
Non-invasive tear break-up time (NITBUT) | 28 days (analysed for each treatment period)
  Measure of time taken from blink to breakup of tear film
Evaporimetry | 28 days (analysed for each treatment period)
  Measure of the rate of evaporation of the tear film from the surface of the eye
Interferometry | 28 days (analysed for each treatment period)
  Tear film lipid layer interferometry is a test to study the structure and quality of the lipid layer in the tear film
Osmolarity | 28 days (analysed for each treatment period)
  Tear osmolarity is a test to determine the solute concentration of the tear film
Corneal and Conjunctival Staining | 28 days (analysed for each treatment period)
  Corneal and conjunctival damage due to dry eye can be measured by staining the surface of the eye with fluorescein and examining under a lamp with a cobalt blue filter
Inflammatory markers | 28 days (analysed for each treatment period)
  Cytokine analysis will be carried out to determine the presence and concentration of a panel of inflammatory biomarkers in the tears using a multiplex immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gupta, Principal Investigator — NHS Greater Glasgow & Clyde

IPD SHARING:
Plan to Share IPD: No